CLINICAL TRIAL: NCT05441553
Title: A Phase 1/2 Study to Evaluate the Safety and Efficacy of VGB-R04 in Adult Hemophilia B Patients
Brief Title: A Study to Evaluate the Safety and Efficacy of VGB-R04 in Adult Hemophilia B Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGB-R04-101
Record Dates: First submitted 2022-06-15; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VGB-R04 (Experimental): Single intravenous (i.v.) infusion of VGB-R04 Intervention: Gene Therapy / Gene Transfer
  Interventions: Genetic: VGB-R04

INTERVENTIONS:
Genetic: VGB-R04 — A novel, bioengineered adeno-associated viral (AAV) vector carrying human factor IX variant

SUMMARY:
A multicenter, open, non-randomized, phase I/II, two-phase clinical study. The dose exploration phase was phase I, and the dose extension phase was phase II.

DETAILED DESCRIPTION:
Hemophilia B is a genetic bleeding disorder caused by pathogenic variants (eg, mutations, deletion) in the FIX gene. HB patients have frequent and potentially life-threatening bleeding and often develop progressive physical disability and pain from chronic haemarthropathy. Current replacement therapy needs regular treatment in the life-long time, bringing heavy economic and social burdens.

VGB-R04 is a novel AAV vector carrying a high specific activity factor IX variant. This study is intended to evaluate the safety, tolerability and efficacy of a single IV infusion of VGB-R04. All subjects in this study will provide informed consent and then undergo screening assessments up to 6 weeks before administration of VGB-R04. All subjects will undergo 52 weeks of safety observation and will be encouraged to enroll in an Long-term follow-up study to evaluate the long-term safety of VGB-R04 for a total of five years.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥18 years and ≤65years of age;
2. Confirmed diagnosis of hemophilia B (baseline FIX activity ≤ 2% of normal);
3. At least 100 days exposure history to FIX;
4. Currently receiving FIX Prophylaxis therapy or on-demand treatment to prevent bleeding;
5. Have acceptable laboratory values:

   1. Hemoglobin ≥110 g/L;
   2. Platelets ≥100×109 /L;
   3. AST, ALT, alkaline phosphatase ≤2×upper limit of normal (ULN) at the testing laboratory;
   4. Bilirubin ≤3× ULN ;
   5. Creatinine ≤1.5× ULN.
6. No measurable factor IX inhibitor as assessed by the central laboratory and have no prior history of inhibitors to factor IX protein;
7. Agree to use reliable contraception until 2 consecutive samples are negative for vector sequences;

Exclusion Criteria:

1. Have significant underlying liver disease within the past 6 months prior to or at Screening, including but not limited to:

   1. Preexisting diagnosis of portal hypertension;
   2. Splenomegaly;
   3. Encephalopathy;
   4. Reduction of serum albumin;
   5. Evidence of significant liver fibrosis;
2. Have anti-VGB-R04 neutralizing antibody titers ≥1:5;
3. Evidence of severe infection disease, i.e., human immunodeficiency virus (HIV) infection, syphilis, tuberculosis, etc.;
4. Novel coronavirus infection occurred in the 6 weeks prior to entry into the group
5. Evidence of active hepatitis B virus infection (HBsAg positive) or hepatitis C virus infection (HCV-RNA positive);
6. Evidence of malignant tumours or those with a previous history of malignant tumours;
7. Have a history of chronic infection or other chronic diseases that the Investigator considers to constitute an unacceptable risk;
8. Any immunodeficiency;
9. planned surgery may be required within one year;
10. Past thromboembolic events (arterial or venous thromboembolic events);
11. Hypertensive patients with poor blood pressure control (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90mmHg after antihypertensive drug treatment);

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Baseline up to Week 52
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
Incidence of serious adverse events | Baseline up to Week 52
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that resulted in death; life threatening;require inpatient hospitalization or prolongation of existing hospitalization; result in persistent or significant disability/incapacity; result in congenital anomaly/birth defect
FIX:C Antigen Level at Steady State | Baseline up to Week 52
  FIX:C activity antigen levels were characterized by post-treatment population mean.

SECONDARY OUTCOMES:
FIX:C activity level | Baseline up to Week 52
  FIX:C activity change from baseline during each visit.
Vector- derived FIX antigen levels | Baseline up to Week 52
  The vector-derived endogenous (not affected by intercurrent FIX product infusions) FIX:C activity antigen levels will be characterized by post-treatment population mean, and its change from baseline during each visit.
Annualized bleeding rate changes from baseline | Baseline up to Week 52
  The annualized numberof bleeding episodes.
Annualized FIX consumption changes from baseline | Baseline up to Week 52
  The annualized use of FIX replacement therapy will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Shanghai Vitalgen Biopharma Co.,Ltd., Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when VGB-R04 is fully approved.
Time Frame: IPD will be shared with other researchers when VGB-R04 is fully approved.
Access Criteria: IPD will be shared with other researchers when VGB-R04 is fully approved.